CLINICAL TRIAL: NCT03864081
Title: Non-Invasive Point-of-care Diagnosis Using Machine Learning and Signal Analytics to Transform Early Detection of Heart Disease
Acronym: IDENTIFY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Analytics For Life (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CADF-CIP-001
Record Dates: First submitted 2019-01-01; First posted 2019-03-06 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary angiography; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Enrolled Subjects (PSR) (Other): Patients who meet the study's inclusion and exclusion criteria, including signing the informed consent form, subjects will undergo signal acquisition prior to their scheduled cardiac catheterization on the day of the procedure.
  Interventions: Device: Phase Signal Recorder

INTERVENTIONS:
Device: Phase Signal Recorder — The Phase Signal Acquisition (PSAQ) System is a medical device system that is being developed to collect phase signals from patients to support the development and testing of machine learned algorithms. The PSAQ System consists of two components that work together to acquire and transmit the phase signals and patient specific data to a secured, cloud-based repository. The PSAQ System is comprised of: 1) the Phase Signal Recorder (PSR) which is a portable instrument, and 2) the Phase Signal Data Repository (PSDR) which is a cloud based data repository. Data collected during this study will not be used to guide treatment.
  Other Names: PSR

SUMMARY:
This study is designed as a repository study to collect resting cardiac phase signals and subject meta data from eligible subjects using the Phase Signal Recorder (PSR) prior to coronary angiography. The repository data will be used for the purposes of research, development, optimization and testing of machine-learning algorithms developed by Analytics 4 Life.

DETAILED DESCRIPTION:
Male and Female subjects will be uniquely and consecutively enrolled into one of two groups to support populating a repository of phase signals: Group 1: Subjects with known prior coronary artery disease or previous percutaneous coronary intervention (PCI), and Group 2: Subjects with new onset symptoms suggestive of obstructive coronary artery disease at current presentation with no known coronary artery disease.

Enrollment into Group 1 and Group 2 will occur simultaneously until up to 500 male subjects and up to 1000 female subjects with paired data (phase signal and coronary angiography outcomes data) are enrolled. Once the desired number of subjects have been enrolled from both groups, then only Group 2 will continue to be enrolled.

Resting phase signals will be collected in all patients who meet inclusion/exclusion criteria and have signed an informed consent form. This study consists of a screening visit, resting phase signal collection (study procedure), and coronary angiography. In this study, resting phase signals will be acquired in subjects prior to coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old;
2. Symptoms suggestive of obstructive CAD;
3. Scheduled to undergo cardiac catheterization with coronary angiography;
4. Ability to understand the requirements of the study and to provide written informed consent.

Exclusion Criteria:

1. Prior documented history of myocardial infarction (MI);
2. Suspected acute myocardial infarction (AMI) at current presentation;
3. Prior coronary artery bypass grafting (CABG);
4. Prior heart valve replacement;
5. Previous sustained or paroxysmal atrial or ventricular arrythmia;
6. Infiltrative myocardial disease (amyloid, sarcoid, right ventricular dysplasia);
7. Presence of cardiac implantable electronic device (CIED), including implantable cardioverter defibrillator (ICD), pacemaker (PM), implantable loop recorders and other monitors;
8. Implantable Neuro-stimulators;
9. Congenital Heart Disease;
10. Pregnant or breast feeding;
11. Currently taking any Type IA, IC or III antiarrhythmics;
12. Any history of amiodarone use;
13. Clinically significant chest deformity (e.g., pectus excavatum or pectus carinatum);
14. Breast implants;
15. Neuromuscular Disease if the condition results in tremor or muscle fasciculations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Phase Signal Recorder Procedure | 7 day
  Resting phase signals will be collected from eligible subjects prior to coronary angiography and paired with angiography results..

CONTACTS AND LOCATIONS:
Overall Officials: William E Sanders, Jr., MD JD LLM MBA FHRS, Study Director — Analytics For Life
Locations (1):
- Atlanta Heart Specialists, Cumming, Georgia, United States

IPD SHARING:
Plan to Share IPD: No